CLINICAL TRIAL: NCT02345902
Title: Randomized Double-Blind Clinical Trial to Compare Haloperidol and Non-Pharmacologic Treatment Versus Non-Pharmacologic Treatment and Placebo, in Elderly Hospitalized Patients With Hypoactive Delirium
Brief Title: Treatment of Hypoactive Delirium and Outcome Measures
Acronym: THDOM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: InstitutoNCMNSZ
Record Dates: First submitted 2014-11-07; First posted 2015-01-26 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2016-01

CONDITIONS: Hypoactive Delirium
MeSH Terms: interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Haloperidol and non-pharmacologic (Experimental): Haloperidol 1.25mg PO q. d. during nine days
  Non-pharmacologic measures:
  A. Reorientation (i.e., calendar, clocks, familiar objects) B. Glasses and hearing devices for the particular patients needing such aids C. Avoidance of physical restraints D. Limitation of excessive personnel shifts or hospital room E. A tranquil and comfortable environment, especially at night, to avoid interruptions (i.e., dim light, low levels of noise) F. Adequate schedules for medication administration and to take vital signs or medical procedures G. Sleep hygiene (light in the room and movement during the day) H. Avoidance of dehydration I. Avoidance of medications use which are associated with delirium (e.g., psychoactive medications)
  Interventions: Drug: Haloperidol; Other: non-pharmacologic measures
- Placebo and non-pharmacologic (Active Comparator): Placebo 1.25 mg PO q.d during nine days.
  Non-pharmacologic measures:
  A. Reorientation (i.e., calendar, clocks, familiar objects) B. Glasses and hearing devices for the particular patients needing such aids C. Avoidance of physical restraints D. Limitation of excessive personnel shifts or hospital room E. A tranquil and comfortable environment, especially at night, to avoid interruptions (i.e., dim light, low levels of noise) F. Adequate schedules for medication administration and to take vital signs or medical procedures G. Sleep hygiene (light in the room and movement during the day) H. Avoidance of dehydration I. Avoidance of medications use which are associated with delirium (e.g., psychoactive medications)
  Interventions: Other: Placebo; Other: non-pharmacologic measures

INTERVENTIONS:
Drug: Haloperidol — haloperidol 1.25 mg P.O q.d
  Other Names: haloperil
  Arms: Haloperidol and non-pharmacologic
Other: Placebo — placebo 1.25 mg P.O q.d
  Arms: Placebo and non-pharmacologic
Other: non-pharmacologic measures — A. Reorientation (i.e., calendar, clocks, familiar objects) B. Glasses and hearing devices for the particular patients needing such aids C. Avoidance of physical restraints D. Limitation of excessive personnel shifts or hospital room E. A tranquil and comfortable environment, especially at night, to avoid interruptions (i.e., dim light, low levels of noise) F. Adequate schedules for medication administration and to take vital signs or medical procedures G. Sleep hygiene (light in the room and movement during the day) H. Avoidance of dehydration I. Avoidance of medications use which are associated with delirium (e.g., psychoactive medications)

SUMMARY:
Haloperidol and Non-Pharmacologic Treatment are recognized treatments for delirium. This study will evaluate which is the best treatment for hypoactive delirium.

DETAILED DESCRIPTION:
Background

Delirium is a cognitive disorder that affects attention and other mental functions. It has an acute onset (in hours or days), a fluctuating course and has various conditioning factors such as diseases or withdrawal or intoxication syndromes.

Delirium is a syndrome with multifactorial origin, it commonly presents in elderly patients, with a prevalence of 20%. Delirium develops when basal vulnerability interacts with precipitating factors.

Delirium has three types according to its psychomotor presentation, hyperactive (agitated), hypoactive (tranquil) or mixed. Delirium has serious outcomes, such as prolonged hospitalization (1), cognitive decline and dementia (2,3,4,), posttraumatic stress disorder (5) and a higher mortality (1).

A neurotransmitter imbalance between acetylcholine and dopamine explains delirium symptoms. A dopamine excess has various consequences: hallucinations that are present in 51 %, and delusions, present in up to 43% in hypoactive delirium. These symptoms produce acute stress in patients and caregivers. It is reported that 53.5% of patients recalled the episode of delirium and from these, 55% of them recalled it associated to hallucinations and 95% of them to delusions. Family recalled the event as stressful in 66%, nurses in 65% of those who did not have hallucinations and in 88% of those who had (6).

Hallucinations and delusions are risk factors for the development of posttraumatic stress disorder, which occurs in up 22% of patients.

Dopamine increase has been associated to apoptosis for its neurotoxic effects. Inflammation has a role in delirium. A study demonstrated that cortisol, Interleukin 6 ( IL-6) and protein S100 calcium binding protein B (S 100β) are all associated with delirium (7).

It is important to note that antipsychotics may have a neuro-protective effect by blocking dopamine receptors, and, therefore, diminishing the potential negative outcomes associated with dopamine excess. Furthermore in an observational study using haloperidol in the intensive care unit there was a decrease in mortality, possibly by its effects on inflammation, inhibiting the release of proinflammatory cytokines (8). One of the effects of haloperidol in vitro is the induction of interleukin receptor antagonist ( IL-IRA), which has shown to have an independent role in delirium. IL-IRA blocks the actions of Interleukin 1α (IL-1α) and interleukin 1β (IL-Iβ) . IL-IRA also downregulates ischaemic and excitotoxic damage (9).

Treatment of Delirium

Psychiatrist, Geriatricians and Neurologists, usually, treat delirium; however treatment strategies vary widely among disciplines, due to differences in the practice guidelines and local applications of current knowledge among centers. An integration of their treatment approaches could offer important clinical advantages. To refer some differences, The American Psychiatric Association (APA) Guidelines (10) recommend treatment with antipsychotics for elderly patients. Where haloperidol is the gold standard, with a dose of 0.25 to 0.50 mg every 4 hours, although the dose may need to be increased for those patients severely agitated. There is no mention among all subtypes of delirium. This guideline recognizes the non-pharmacologic intervention as part of the treatment.

On the other hand, Geriatrics Guidelines for the treatment of delirium, mention that the treatment of delirium should be mainly based on non-pharmacologic treatment. Restricting the pharmacologic treatment for those patients with severe manifestations of agitation (11). The NICE Guidelines mention that pharmacologic treatment in hypoactive delirium patients is indicated during one week to those patients with distress due to hallucinations (12).

Authors have mentioned that non-pharmacologic measures have not been assessed in clinical trials, and that pharmacologic treatment has not been recommended at this time (13). Furthermore, others addressed that currently, treatment with antipsychotics are used where non-pharmacologic measures have failed to treat psychotic symptoms. Or when the safety of patients or others are compromised, and that clinical trials with antipsychotics are few (14).

As it was mentioned before, there is no standardized treatment of delirium among different disciplines. Therefore, it is still on debate to determine which the best strategy in treating delirium is.

As far as we know, there are no clinical trials adequately evaluating haloperidol as the cornerstone of management in hypoactive delirium. Nonetheless, those patients who were exposed to a higher dose of haloperidol improved significantly with this antipsychotic (15).

Therefore, it is not known whether hypoactive delirium (the most frequent and difficult to recognize) should be treated with haloperidol at lower doses. Or if haloperidol should be used only in mixed and hyperactive types of delirium. Though despite few studies that have included patients with hypoactive delirium suggest that antipsychotics may have a role in the treatment of this delirium subtype (16).

Statement of the Problem

Hypoactive delirium is a common condition in hospitalized elderly patients. It is the most common type of delirium that carries more difficulty in its diagnosis. It is associated to a longer hospital stay, increased expenses associated to its diagnosis and more doubts on the most efficacious treatment strategy.

Surprisingly, even when hypoactive delirium is the most frequent, it is the hyperactive type the paradigm of study, and it is the one specifically mentioned in treatment guidelines.

To the best of our knowledge, there are no studies evaluating specifically haloperidol in hypoactive delirium. Some studies have excluded this type of delirium systematically or include all delirium subtypes where hypoactive delirium is poorly represented/analyzed.

Significance of the Investigation

There are few clinical studies correctly designed, exempt of methodological flaws and evaluating the most important clinical outcomes in delirium patients in general. There are no randomized clinical trials (RCTs) testing low-dose haloperidol against non-pharmacologic measures in the treatment of hypoactive delirium. Just few studies have included patients with hypoactive delirium with varying results, contributing to the lack of uniform recommendations (16). Currently, its treatment is based on the particular experiences of each clinical center without measuring its impact on relevant outcomes.

Furthermore, there are no studies evaluating perceived stress in patients and their caregivers, as well as posttraumatic stress in hypoactive delirium patients. None has evaluated cognitive decline after a hypoactive delirium treated either with antipsychotics or non-pharmacologic measures.

The purpose of the present RCT is to bring out knowledge about different treatments in elderly patients with hypoactive delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill criteria for delirium according to CAM and DOSS
* Patients in hospitalization who are not receiving treatment for delirium
* Patients without treatment with antipsychotics for any other reason
* Patients whose legally proxy accepts to participate

Exclusion Criteria:

* Patients who have received pharmacologic treatment for delirium
* Patients with a corrected QT interval prolongation
* Patients who receive antipsychotics for any other reason
* Patients in another age group
* Patients whose legally proxy does not accept to participate
* Patients with dementia
* Patients with Parkinson disease
* Patients with arrythmias
* Patients with language or hearing disorders that impede communication
* Patients hospitalized in the Intensive Care Unit
* Patients who are receiving benzodiazepines and anticholinergics
* Patients with dopamine agonists or antagonists
* Patients who develop a severe neurologic disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in delirium severity | Participants will be followed at an expected average of nine days
  Reduction of 50% from the basal DOSS score

SECONDARY OUTCOMES:
Necessity of additional open label haloperidol doses to control delirium symptoms | Participants will be followed at an expected average of nine days
  In case the patient develops a hyperactive state will receive haloperidol in an open label dose, 1 mg that could be repeated every 4 hours in case the agitation persists, for a maximum daily dose of 6 mg. In this way, the dose will never exceed the recommended 10 mg dose per day.
  If the patient persists with a hypoactive state (absence of improvement on the DOSS score), we will increase the dose to 2.5 mg or half a tablet (of haloperidol or placebo q.d.) or 3.75 mg,three quarters of a tablet ( of haloperidol or placebo q.d.)
Delirium duration | Participants will be followed at an expected average of nine days
  Using the DOSS basal score and the CAM
Perceived stress | At 24 hours after delirium remission
  in patients, health staff and caregivers of both groups using the delirium experience questionnaire
Posttraumatic stress disorder | At 6 months after delirium remission
  In patients of both groups using the posttraumatic stress disorder section of the Mini International Neuropsychiatry Interview
Cognitive impairment as assessed by Montreal Cognitive Assessment (MoCA) <24 points | At 6 months after delirium remission
  Number of patients with <24 points in the Montreal Cognitive Assessment at 6 months after delirium remission, as compared with the number of patients with scoring >3.5 points in the Informant Questionnaire on Cognitive Decline in the Elderly, as an estimate of the baseline (pre-delirium) state
Cerebral blood flow as assessed by transcranial Doppler | At baseline and after 24 h of delirium remission
  in patients of both groups using a cerebral ultrasound
Side effects associated with either intervention | Participants will be followed at an expected average of nine days
  We will list all adverse reactions associated with haloperidol (extra pyramidal effects, arrhythmias, hypersensitivity to the drug or corrected QT interval prolongation), the medication will be stopped in case of the appearance of an life-threatening reaction. We will consider this case when a patient needs ventilator support, use of cardiac amines, hemodialysis or the use of the Intensive Care Unit. These conditions will require opening the masking and exit the patient from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Erwin Chiquete, MD, PhD, Study Director — Instituto Nacional de Ciencias Médicas y Nutrición; Carlos Cantú, MD, PhD, Study Director — Instituto Nacional de Ciencias Médicas y Nutrición
Locations (1):
- Department of Neurology and Psychiatry. Instituto Nacional de Ciencias Médicas y Nutrición, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khan BA, Zawahiri M, Campbell NL, Fox GC, Weinstein EJ, Nazir A, Farber MO, Buckley JD, Maclullich A, Boustani MA. Delirium in hospitalized patients: implications of current evidence on clinical practice and future avenues for research--a systematic evidence review. J Hosp Med. 2012 Sep;7(7):580-9. doi: 10.1002/jhm.1949. Epub 2012 Jun 8. PMID 22684893
- [Background] McCusker J, Cole M, Dendukuri N, Belzile E, Primeau F. Delirium in older medical inpatients and subsequent cognitive and functional status: a prospective study. CMAJ. 2001 Sep 4;165(5):575-83. PMID 11563209
- [Background] Davis DH, Muniz Terrera G, Keage H, Rahkonen T, Oinas M, Matthews FE, Cunningham C, Polvikoski T, Sulkava R, MacLullich AM, Brayne C. Delirium is a strong risk factor for dementia in the oldest-old: a population-based cohort study. Brain. 2012 Sep;135(Pt 9):2809-16. doi: 10.1093/brain/aws190. Epub 2012 Aug 9. PMID 22879644
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Griffiths RD, Jones C. Delirium, cognitive dysfunction and posttraumatic stress disorder. Curr Opin Anaesthesiol. 2007 Apr;20(2):124-9. doi: 10.1097/ACO.0b013e3280803d4b. PMID 17413395
- [Background] Breitbart W, Gibson C, Tremblay A. The delirium experience: delirium recall and delirium-related distress in hospitalized patients with cancer, their spouses/caregivers, and their nurses. Psychosomatics. 2002 May-Jun;43(3):183-94. doi: 10.1176/appi.psy.43.3.183. PMID 12075033
- [Background] van Munster BC, Bisschop PH, Zwinderman AH, Korevaar JC, Endert E, Wiersinga WJ, van Oosten HE, Goslings JC, de Rooij SE. Cortisol, interleukins and S100B in delirium in the elderly. Brain Cogn. 2010 Oct;74(1):18-23. doi: 10.1016/j.bandc.2010.05.010. Epub 2010 Jun 26. PMID 20580479
- [Background] Milbrandt EB, Kersten A, Kong L, Weissfeld LA, Clermont G, Fink MP, Angus DC. Haloperidol use is associated with lower hospital mortality in mechanically ventilated patients. Crit Care Med. 2005 Jan;33(1):226-9; discussion 263-5. doi: 10.1097/01.ccm.0000150743.16005.9a. PMID 15644675
- [Background] Adamis D, Lunn M, Martin FC, Treloar A, Gregson N, Hamilton G, Macdonald AJ. Cytokines and IGF-I in delirious and non-delirious acutely ill older medical inpatients. Age Ageing. 2009 May;38(3):326-32; discussion 251. doi: 10.1093/ageing/afp014. Epub 2009 Mar 5. PMID 19269948
- [Background] Practice guideline for the treatment of patients with delirium. American Psychiatric Association. Am J Psychiatry. 1999 May;156(5 Suppl):1-20. No abstract available. PMID 10327941
- [Background] Brajtman S, Wright D, Hogan DB, Allard P, Bruto V, Burne D, Gage L, Gagnon PR, Sadowski CA, Helsdingen S, Wilson K. Developing guidelines on the assessment and treatment of delirium in older adults at the end of life. Can Geriatr J. 2011 Jun;14(2):40-50. doi: 10.5770/cgj.v14i2.13. Epub 2011 Jul 7. PMID 23251311
- [Background] National Clinical Guideline Centre (UK). Delirium: Diagnosis, Prevention and Management [Internet]. London: Royal College of Physicians (UK); 2010 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK65558/ PMID 22319805
- [Background] Inouye SK, Westendorp RG, Saczynski JS, Kimchi EY, Cleinman AA. Delirium in elderly people--authors'reply. Lancet. 2014 Jun 14;383(9934):2045. doi: 10.1016/S0140-6736(14)60994-6. No abstract available. PMID 24931690
- [Background] Maclullich AM, Anand A, Davis DH, Jackson T, Barugh AJ, Hall RJ, Ferguson KJ, Meagher DJ, Cunningham C. New horizons in the pathogenesis, assessment and management of delirium. Age Ageing. 2013 Nov;42(6):667-74. doi: 10.1093/ageing/aft148. Epub 2013 Sep 25. PMID 24067500
- [Background] Boettger S, Friedlander M, Breitbart W, Passik S. Aripiprazole and haloperidol in the treatment of delirium. Aust N Z J Psychiatry. 2011 Jun;45(6):477-82. doi: 10.3109/00048674.2011.543411. PMID 21563866
- [Background] Friedman JI, Soleimani L, McGonigle DP, Egol C, Silverstein JH. Pharmacological treatments of non-substance-withdrawal delirium: a systematic review of prospective trials. Am J Psychiatry. 2014 Feb;171(2):151-9. doi: 10.1176/appi.ajp.2013.13040458. PMID 24362367